CLINICAL TRIAL: NCT01618773
Title: Epiduo in the Long-term Treatment of Moderate to Severe Acne With or Without Concomitant Medication
Brief Title: Long-term Study of Epiduo in Patients With Moderate to Severe Acne
Acronym: ELANG
Status: Completed | Type: Observational
Sponsor: Galderma Laboratorium GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: ELANG
Record Dates: First submitted 2012-06-12; First posted 2012-06-13 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Acne Vulgaris
Keywords: acne; Epiduo; adapalene/ benzoyl peroxide
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Benzoyl Peroxide; Adapalene, Benzoyl Peroxide Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 0.1% adapalene / 2.5% benzoyl peroxide — topical application
  Other Names: Epiduo

SUMMARY:
This observational study is designed to assess the long-term efficacy and safety of Epiduo (alone or in combination with other drugs) under daily clinical practice conditions in patients with moderate to severe inflammatory acne. In addition, the effect of Epiduo on quality of life and patient adherence will be assessed under marketed conditions.

DETAILED DESCRIPTION:
This observational study is designed to assess the long-term efficacy and safety of Epiduo under daily clinical practice conditions. The study includes patients of all ages with moderate to severe inflammatory acne, taking Epiduo alone or in combination with other drugs. In addition, the effect of Epiduo alone or in combination with other drugs on quality of life and patient adherence will be assessed under marketed conditions.

The observational study is designed as a multicentre study, covering all parts of Germany. Participating investigators are dermatologists with an adequate patient pool of acne patients. The observation time per patient will be 9 months. An interim and final examination with subsequent documentation are designated to be performed about 3 and 9 months after the start of treatment, respectively.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been diagnosed with moderate to severe inflammatory acne (Leeds Grade 4-12)
* Topical therapy of acne with Epiduo is indicated, the decision about treating the patient with Epiduo has been made independently from this study

Exclusion Criteria:

* Use of Epiduo within 3 months prior to inclusion
* Pregnancy or breastfeeding
* Acne inversa
* Acne with preferential manifestation of microcysts, macrocysts and macrocomedones
* Hypersensitivity to the drug or any of its ingredients
* If applicable, other restrictions outlined in the SPC of Epiduo

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: About 6,650 patients with moderate to severe acne (Leeds grade 4-12)
Sampling Method: Probability Sample
Enrollment: 6036 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Severity of acne | at baseline and after 3 and 9 months treatment
  Efficacy is assessed by change in severity of acne according to the Leeds revised grading system

SECONDARY OUTCOMES:
Quality of Life | at baseline and after 3 and 9 months of treatment
  Quality of life is assessed using the Cardiff Acne Disability Index
Treatment adherence | after 3 and 9 months of treatment
  Treatment adherence is assessed by the physician using a mini-questionnaire published by the international acne expert group "Global Alliance to Improve Outcomes in Acne"
Local Skin Irritations | over 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Harald PM Gollnick, Prof. Dr., Principal Investigator — Universitätsklinikum Magdeburg A.ö.R. Klinik für Dermatologie und Venerologie

IPD SHARING:
Plan to Share IPD: No